CLINICAL TRIAL: NCT04372849
Title: Insulinsensitivität Des Menschlichen Zentralnervensystems Mit Fortschreitendem Alter: Kernspintomographische Untersuchung Mit Intranasaler Gabe Von Insulin
Brief Title: Effects of Age and Obesity on Brain Insulin Sensitivity
Acronym: Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 837/2016BO2
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-04

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal insulin spray (Active Comparator)
  Interventions: Other: Human nasal insulin
- Placebo spray (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Human nasal insulin — single dose of 160 U of human insulin as nasal spray
  Arms: Nasal insulin spray
Other: Placebo — Single dose of placebo solution as nasal spray
  Arms: Placebo spray

SUMMARY:
Obesity and especially type 2 diabetes (T2D) increases the risk of neurocognitive dysfunctions including adverse effects on brain structure and function. Recent evidence from clinical studies have shown that T2D almost doubles the risk for dementia. As the population gets older, age-related chronic diseases, as T2D, become more prevalent. Scientific evidence is emerging that there are several links between metabolic and neurocognitive functions. Impaired insulin action (i.e. insulin resistance), the main hallmark of T2D, has been suggested as a likely shared common pathophysiological mechanism. However, the neural processes that determine how insulin resistance is are connected to the onset and progression of T2D and dementia remain unclear. In this context, the overall aim is to study brain insulin resistance to disentangle age-related and obesity related brain insulin resistance in healthy normal and overweight/obese persons at the age of 20 to 70 years . To this end, the investigators will assess brain insulin action using intranasal insulin/placebo during functional Magnetic Resonance Imaging (fMRI). Additionally, structural changes and cognitive processes will be assessed as secondary variables.

ELIGIBILITY:
Inclusion Criteria:

* Body-Mass Index (BMI) between 19-35 kg/m2
* HbA1c ≤6.0%
* normal glucose tolerance during 75g oral glucose tolerance test (OGTT)

Exclusion Criteria:

* Not removable metal parts in or on the body
* manifest cardiovascular disease
* claustrophobia
* recent surgery (less than 3 months)
* Simultaneous participation in other studies
* Acute disease or infection within the last 4 weeks
* neurological and psychiatric disorders
* treatment with centrally acting drugs
* hemoglobin Hb <13g / dl
* Hypersensitivity to any of the substances used

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Brain insulin sensitivity in different age,weight and sex groups | 30 minutes after administration of nasal insulin
  fMRI measurement will be performed before and after administration of 160 U of human insulin or placebo as nasal spray. Changes in regional brain activity will be quantified by cerebral blood flow and blood oxygenation dependent (BOLD) signal to assess regional brain insulin sensitivity. Brain insulin sensitivity will be compared between eight groups (young normal weight men and women, young overweight/obese men and women, old normal weight men and women, old overweight/obese men and women). Persons are categorized into normal weight and overweight/obese based on the Body Mass Index (BMI). Age groups are build based on a median split.

SECONDARY OUTCOMES:
Whole-body insulin sensitivity | 2 hours
  Insulin sensitivity will be estimated from a frequent-sampling 75 g oral glucose tolerance test (oGTT) using the Matsuda formula. Correlation of regional brain insulin sensitivity by intranasal insulin will be performed with whole-body insulin sensitivity based on oGTT. Changes in regional cerebral blood flow from before to after intranasal insulin administration will be assessed by functional magnetic resonance imaging (fMRI).
Correlation with autonomous nervous system activity | 10 - 150 minutes post nasal spray
  Correlation of the change in regional brain insulin sensitivity by intranasal insulin with the simultaneous change of the autonomous nervous system (measured by heart rate variability).
Correlation with cognitive function | 1 hours
  Correlation of the change in regional brain insulin sensitivity by intranasal insulin with cognitive measures addressed by neuropsychological testing.
Response to food cues | 20 minutes
  Brain response to food cues assessed by functional magnetic resonance imaging. Food cues will be rated for palatability on a visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany